CLINICAL TRIAL: NCT00468585
Title: A Multicenter, Phase I/II Study of Every Other Week Capecitabine Dosing With Bevacizumab for the Treatment of Metastatic Breast Cancer Based Upon the Norton-Simon Mathematical Model
Brief Title: Study of Biweekly Capecitabine Dosing With Bevacizumab for the Treatment of Metastatic Breast Cancer Based Upon the Norton-Simon Mathematical Model
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-030
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metastatic breast cancer; Breast; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Capecitabine and Bevacizumab (Experimental): The Phase II trial has a Simon mini-max two-stage design. Twenty-seven patients will be enrolled to the first stage of the Phase II trial, with a target accrual of 40 patients. The treatment dose of capecitabine as determined in the Phase I portion of this trial will be administered orally in two divided doses daily on Days 1 through 7 and Days 15 through 21 in a 28 day cycle. Phase II patients will receive bevacizumab 10 mg/kg intravenously every 2 weeks concurrently with oral capecitabine. Patients will be evaluated for toxicity between Days 3 to 5 (complete blood count only), Day 8, Day 15, and Day 22 during cycle #1. Thereafter, toxicity will be assessed on Days 1 and 15. Efficacy will be assessed with every other week physical examination and radiographic scans of measurable disease every 12 weeks.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine
Drug: Bevacizumab

SUMMARY:
The purpose of this study is to find out what effects (both good and bad) that capecitabine has on you and your breast cancer when given in a novel schedule in combination with the antibody therapy, bevacizumab. Capecitabine (Xeloda®) is an anticancer drug that was approved by FDA in 1998 for treating metastatic breast cancer. Capecitabine is a pill that blocks the way cancer cells multiply and grow. Usually, this medicine is taken twice a day for fourteen days in a row.

Patients then get a break from the drug for seven days. With this schedule and usual dose, some patients on capecitabine have experienced side effects that interfered with their daily comfort.Different doses and schedules of capecitabine have been studied in animal studies and in people with colon cancer. Mathematic modeling has been used to better understand these results.Information from these experiments leads us to ask if 7 days of treatment with capecitabine followed by a 7-day break is both safer and more active against breast cancer. The study you are considering is a first step in this direction and is designed to demonstrate both safety and activity.

Bevacizumab is a biologic therapy that targets the growth of blood vessels which tumors need to grow. Women whose breast cancer spread to other parts of their bodies lived longer without their cancers growing when they were treated with bevacizumab and chemotherapy. Bevacizumab was tested with the 14-day/7-day schedule of capecitabine. These two medicines are safe when given together and seem to work better against breast cancer than capecitabine alone.

This study is designed to answer the questions:

1. What are the side effects of bevacizumab and capecitabine when given in this different schedule and how often do they occur?
2. When given in this schedule, does capecitabine with bevacizumab help treat breast cancer that has spread or continues to grow despite being treated by other chemotherapy drugs before?

DETAILED DESCRIPTION:
A. Primary Objectives:

• To estimate the efficacy of every other week capecitabine and bevacizumab in patients with metastatic breast cancer in terms of overall response rate (complete response (CR) + partial response (PR)) when administered at the MTD of capecitabine determined by the phase I portion of this trial.

B. Secondary Objectives:

* To estimate secondary efficacy endpoints of this combination including clinical benefit (CR+PR+SD > 6 months), time to tumor progression (TTP), progression free survival (TTP) and duration of response.
* To evaluate toxicity rates associated with this capecitabine schedule in combination with bevacizumab using the NCI CTC (version 3) and the Hand-Foot Syndrome Grading Scale developed by Roche Laboratories, Inc.
* To evaluate the pharmacogenetics of capecitabine in breast cancer patients by assessing the impact of specific candidate SNPs on toxicity and/or response.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) with diagnosis of invasive adenocarcinoma of the breast confirmed at MSKCC either by histology or cytology.
* Clinical evidence of metastatic breast cancer, non-amenable to surgery or radiation therapy with curative intent.
* Presence of at least one measurable metastatic lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable. Minimum indicator lesion size: greater than or equal to 10 mm measured by spiral CT or greater than or equal to 20 mm measured by conventional techniques.
* Any number of prior endocrine or biologic therapies is permitted on this trial. In addition, patients may be untreated in the metastatic setting or have received any number of prior cytotoxic regimens. All previous chemotherapy must have been discontinued at least 3 weeks prior to study entry. All acute toxic effects (excluding alopecia or neurotoxicity) of any prior therapy must have resolved to NCI CTC (Version 3) Grade less than or equal to 1.
* Endocrine therapy with an aromatase inhibitor, SERM (ie, tamoxifen) or fulvestrant is permitted within 4 weeks of study entry, however concurrent therapy with these drugs is not acceptable.
* ECOG performance status of 0, 1 or 2.
* Patients must be either HER2-negative or HER2-positive and no longer a candidate for trastuzumab therapy. HER2-negative is defined as 0 or 1+ staining on immunohistochemistry or FISH negative for gene amplification. HER2-positive is defined as 3+ staining on immunohistochemistry or FISH positive for gene amplification.
* Age greater than or equal to 18 years old.
* Baseline laboratory data within the following limits:
* Absolute neutrophil count (ANC) >1.5 x 10^9/L
* Platelets > 100 x 10^9/L
* Estimated creatinine clearance greater than or equal to 50 ml/min by - Cockcroft-Gault equation
* Total serum bilirubin <1.5 x upper normal limit
* ALT, AST < 2.5x upper normal limit (or <5x upper normal limit in the case of liver metastases)
* Alkaline phosphatase < 2.5x upper normal limit (or >5x upper normal limit in the case of liver metastases or >10x upper normal limit in the case of bone disease)
* Serum or urine pregnancy test for females of childbearing potential Negative within 14 days of starting treatment

Exclusion Criteria:

* Pregnant or nursing women may not participate. Patients of reproductive potential may not participate unless they have agreed to use an effective method of contraception and to continue contraception for 30 days from the date of the last study drug administration. Postmenopausal woman must be amenorrheic for at least 12 months to be considered of nonchildbearing potential.
* Life expectancy < 3 months.
* Serious, uncontrolled, concurrent infection.
* Any prior fluoropyrimidine therapy with the exception of adjuvant administration. Adjuvant fluoropyrimidine containing therapy must be completed at least 6 months prior to enrollment.
* Prior severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil. A history of DPD deficiency will exclude patients from the trial.
* Completion of previous chemotherapy regimen <3 weeks prior to the start of study treatment.
* Prior adjuvant hormonal therapy is permitted. Use of an aromatase inhibitor, anti-estrogen or fulvestrant must be discontinued prior to treatment start.
* Biologic therapy (eg, bevacizumab,trastuzumab) for the treatment of metastatic disease must be discontinued >3 weeks from the start of protocol treatment.
* HER2-positive patients who are candidates for treatment with trastuzumab are excluded from this trial as the concurrent use of trastuzumab may confound study results.
* History of prior malignancy with the following exceptions: adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission (with no evidence of disease) for more than five years.
* Non-malignant systemic disease (cardiovascular, renal, hepatic etc) that would preclude any of the study therapy drugs. Specifically excluded are the following cardiac conditions:

  * Inadequately controlled hypertension (defined as blood pressure of >150/100 mmHg on antihypertensive medications)
  * Any prior history of hypertensive crisis or hypertensive encephalopathy
  * New York Heart Association (NYHA) Class II or greater congestive heart failure
  * History of myocardial infarction or unstable angina within 6 months
  * History of stroke or transient ischemic attack within 6 months
  * Significant vascular disease or symptomatic peripheral vascular disease
* Capecitabine is contraindicated in patients with a creatinine clearance of <30 ml/min.Patients with a creatinine clearance less than 50 ml/minute by Cockroft and Gault Equation will be excluded from the trial.
* Patients with symptomatic CNS metastases that remain untreated by radiation therapy are excluded from this trial. The presence of asymptomatic brain metastases or brain metastases that have been previously irradiated are not grounds for trial exclusion for the phase I study however, these patients are excluded from the phase II portion of the trial.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Other severe, acute or chronic, medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results. Any of the above criteria that in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Presence of uncontrolled gastrointestinal malabsorption syndrome.
* Concurrent use of oral warfarin anticoagulant therapy is not permitted due to serious drug interactions with capecitabine. Full dose anticoagulation with low molecular weight heparin or other (non-warfarin) anticoagulant is permitted.
* Unwillingness to give written informed consent or unwillingness to participate or inability to comply with the protocol for the duration of the study. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures are necessary for participation in this clinical trial.
* Concurrent radiation therapy is not permitted during treatment on protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Related Info — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 0: Capecitabine - AM 1500mg; PM 1500 mg; total daily 3000 mg
- Group 1: Capecitabine - AM 1500 mg; PM 2000 mg; total daily 3500 mg
- Group 2: Capecitabine - AM 2000 mg; PM 2000 mg; total daily 4000 mg
- Group 3: Capecitabine - AM 2000 mg; PM 2500mg; total daily 4500 mg
Period: Overall Study
Arm/Group | Group 0 | Group 1 | Group 2 | Group 3
Started | 4 | 3 | 50 | 6
Completed | 3 | 3 | 45 | 5
Not Completed | 1 | 0 | 5 | 1
Not completed — Patient not treated | 1 | 0 | 1 | 0
Not completed — Patient found to be ineligible | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 0 | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 4 | 3 | 50 | 6 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 46 | 6 | 59
  >=65 years | 0 | 0 | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 50 | 6 | 63
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: This is defined as the percentage of patients who achieve either an objective complete or partial target lesion response that is confirmed based on the RECIST criteria.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Group 0 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 3 | 3 | 45 | 5
participants
  Partial Response (PR) | 0 | 0 | 8 | 0
  Stable Disease (SD) | 2 | 1 | 22 | 3
  Progression of Disease (POD) | 1 | 2 | 15 | 2

ADVERSE EVENTS:
Arm/Group | Group 0 | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 7/50 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 41/50 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 0 (N=4) | Group 1 (N=3) | Group 2 (N=50) | Group 3 (N=6)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Back (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 0 (N=4) | Group 1 (N=3) | Group 2 (N=50) | Group 3 (N=6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
ALT, SGPT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
AST, SGOT (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 10 (10) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 2 (2) | 7 (7) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 14 (14) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Hot flashes/flushes (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Infection, other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 7 (7) | 0 (0)
Pain - Back (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain - Chest wall (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain - Extremity-limb (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Head/headache (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pain - Other (General disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 28 (28) | 3 (3)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (fainting) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes